CLINICAL TRIAL: NCT06153992
Title: Clinical Application of Portable Intelligent Multi Joint Isokinetic Training and Evaluation System Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ran Shi (Other)
Responsible Party: Sponsor-Investigator, Ran Shi, doctor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021004
Record Dates: First submitted 2022-11-04; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Hemiplegia; Rehabilitation; Tobacco Use; Physical Disability
MeSH Terms: conditions — Stroke; Hemiplegia; Tobacco Use

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): The control group received exercise therapy (once a day, 40min/ times, 5 times/week), occupational therapy (once a day, 30min/ times, 5 times/week), low-frequency electricity (once a day, 20min/ times, 5 times/week), acupuncture therapy (once a day, 20min/ times, 5 times/week) .
  Interventions: Other: without test training
- Traditional isokinetic treatment group (Active Comparator): The treatment machine adopts the traditional isokinetic training machine, the treatment items and the treatment parameters are the same as the intelligent isokinetic treatment group.
  Interventions: Device: isokinetic muscle strength test training; Other: without test training
- Intelligent isokinetic treatment group (Experimental): In the intelligent isokinetic treatment group, isokinetic muscle strength training of hemiplegic lower limb flexion muscle group and knee extension muscle group was added to the treatment of the control group.
  Intelligent isokinetic treatment to increase the above treatment hemiplegic lower limb flexion, knee extension muscle isokinetic strength training. The patient's seat back was adjusted to 85° and fixed with a belt and shoulder cross-strap. The thigh of the subject was fixed with a nylon buckle, the lateral condyle of the femur was the axis, the lever arm length was scale 12, and the distal leg was fixed above the ankle. Passive joint activities were performed on the knee and ankle before training. Avoid joint damage and perform three low-resistance warm-up exercises. Choose 60°/s, 90°/s, 120°/s angular speed isokinetic training according to the patient's specific conditions. Each angular speed training is 10 times, the interval rest is 15s.ect.
  Interventions: Device: Intelligent portable isokinetic muscle strength test training; Other: without test training

INTERVENTIONS:
Device: Intelligent portable isokinetic muscle strength test training — The isokinetic training of knee flexors and extensors was carried out by using intelligent portable isokinetic muscle strength test training system
  Arms: Intelligent isokinetic treatment group
Device: isokinetic muscle strength test training — The isokinetic training of knee flexors and extensors was carried out by using isokinetic muscle strength test training system
  Arms: Traditional isokinetic treatment group
Other: without test training — Treatment was performed without using any isokinetic muscle strength test training system

SUMMARY:
The goal of this clinical trial is to compare in describeparticipant population. The main question it aims to answer is:By using intelligent portable isokinetic tester and traditional isokinetic tester, isokinetic knee flexor and extensor muscles of stroke patients with hemiplegia were trained respectively, so as to observe and compare the effects of the two treatment methods. In addition, the therapeutic effect of the above two treatments was compared with that of exercise therapy alone. Participants will be divided into three groups: control group, intelligent isokinetic treatment group, and traditional isokinetic treatment group. Participants of both the control group and the two treatment groups received exercise therapy. On the basis of exercise therapy, participants of the intelligent isokinetic treatment group used the intelligent portable isokinetic tester to train the affected knee flexion and extensor muscle, while the participants of traditional isokinetic treatment group used the intelligent portable isokinetic tester to train the affected knee flexion and extensor muscle.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Cerebral apoplexy's Disease
* Confirmed by CT or MR Examination of the head
* First onset, duration ≤1 month
* The lower extremity of the hemiplegic limb was above Brunnstrom stage III
* Must be able to sign the informed consent form

Exclusion Criteria:

* Vital signs are unstable
* Severe cognitive, visual and hearing impairment
* Orthopaedic disease
* Muscle pain lower extremity
* Congenital disease
* History of other encephalopathy
* History of mental illness

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Body function | up to 1 month
  Evaluate lower limb motor function using the Fugl Meyer method (total lower limb motor score 0-34 points, total balance score 0-14 points).
Measured peak moment | up to 1 month
  Peak moment of knee joint at 60 °/s angular velocity in Nm

SECONDARY OUTCOMES:
Satisfaction questionnaire survey | up to 1 month
  Survey of patients' comfort and satisfaction with the treatment process and effectiveness(score 0-100 points).

CONTACTS AND LOCATIONS:
Overall Officials: Sanyuan Hu, doctor, Study Chair — Qianfoshan Hospital
Locations (1):
- Intelligent Multi Joint Isokinetic, Jinan, Shandong, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT06153992/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT06153992/ICF_001.pdf